CLINICAL TRIAL: NCT05245370
Title: Social Learning Trial: Using Patient and Clinician Testimonials to Modify Treatment Expectations and Placebo Treatments in Depression
Brief Title: Modifying Treatment Expectations in Depression: the Role of Social Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Winfried Rief, Professor, Dr., Philipps University Marburg
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: Social learning_testimonials
Record Dates: First submitted 2022-01-22; First posted 2022-02-17 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Health Care Utilization
Keywords: treatment expectations; social learning; psychotherapy; depression; testimonials
MeSH Terms: conditions — Patient Acceptance of Health Care; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control group 1: Control video (Active Comparator)
  Interventions: Behavioral: Control video
- Control group 2: Rationale video + control video (Active Comparator)
  Interventions: Behavioral: Control video; Behavioral: Rationale video
- Rationale video + clinician testimonial (Experimental)
  Interventions: Behavioral: Rationale video; Behavioral: Clinician testimonial
- Rationale video + patient testimonial (Experimental)
  Interventions: Behavioral: Rationale video; Behavioral: Patient testimonial
- Rationale video + clinician testimonial + patient testimonial (Experimental)
  Interventions: Behavioral: Rationale video; Behavioral: Clinician testimonial; Behavioral: Patient testimonial

INTERVENTIONS:
Behavioral: Control video — Control group 1 will see a control video consisting of basic information about the different types of psychotherapy that are covered by insurance in Germany and the process of applying for psychotherapy with the insurance. The control video is matched in duration (10 minutes), set-up and the overall topic (psychotherapy) to the intervention video testimonials.
  Arms: Control group 1: Control video; Control group 2: Rationale video + control video
Behavioral: Rationale video — The active control group 2 will see a short rationale and the control video. The rationale is a 2:45 minute-long animated video (designed via the visual communication platform powtoon, https://powtoon.com/) explaining some of the underlying mechanisms of depression.
  Arms: Control group 2: Rationale video + control video; Rationale video + clinician testimonial; Rationale video + clinician testimonial + patient testimonial; Rationale video + patient testimonial
Behavioral: Clinician testimonial — This group will see the rationale video first, followed by testimonial of a professional clinician/psychotherapist.
  Arms: Rationale video + clinician testimonial; Rationale video + clinician testimonial + patient testimonial
Behavioral: Patient testimonial — This group will see the rationale video first, followed by testimonial of a patient who is being treated for depression with psychotherapy.
  Arms: Rationale video + clinician testimonial + patient testimonial; Rationale video + patient testimonial

SUMMARY:
Research has shown that treatment expectations play a major role in the course of mental disorders and that positive expectations have a beneficial impact on treatment outcomes. Expectations can develop in different ways, whereby an emerging body of research has shown that social learning plays a significant role in this process. To date, most studies have investigated the impact of social learning on treatment expectations in the context of pain relief. Little is known about the impact of social learning in the psychotherapeutic treatment of depression. Therefore, this study investigates whether treatment expectations regarding the treatment of depression can be modulated via social learning, i.e., showing positive treatment testimonials.

Hypotheses:

H1: The investigators predict that individuals who are provided with treatment testimonials (experimental groups) show a greater change toward positive treatment expectations compared to individuals who do not view such testimonials (control groups).

H2: The investigators predict that individuals provided with treatment testimonials will, compared to the control groups, show a greater change in secondary outcome variables in the following ways: a greater decrease in perceived uncertainty/ barriers; a greater decrease in stigma/ negative attitudes toward psychotherapy; a greater increase in intentions to seek therapy; a greater willingness to try the specific technique described in the videos.

H3: Inter-individual differences in the effect of provided testimonials are associated with pre-existing factors: level of depressive symptoms; intolerance of uncertainty; treatment experience; locus of control; general self-efficacy; dispositional optimism and cognitive immunization tendencies.

Exploratory questions:

1. An exploratory aim of this study is to assess whether viewing different types of testimonials (clinician delivered; patient-delivered; combination of both) has differential effects on treatment expectation change.
2. Furthermore, the investigators want to assess whether implicit treatment expectations change in a similar pattern as explicit treatment expectations.
3. Based on the results of H1 and H2, the investigators aim to assess possible mechanisms of change: e.g. assess whether a change in treatment expectations is mediated by a decrease in perceived uncertainty or a change in stigma/ attitudes toward therapy.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* be able understand German (at least B1 level)
* have access to a computer device with internet access

Exclusion Criteria:

* age below 18 years old
* non correctable hearing or visual impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in scores on the Credibility and Expectancy Questionnaire (CEQ) scale | Baseline; post-Intervention (1 day after baseline, after viewing the intervention videos)
  German version of the Credibility and Expectancy Questionnaire (CEQ), 6-item scale (Raeke, 2013).The CEQ consists of two subscales with four items measuring cognitive-focused credibility (e.g., "At this point, how logical does the therapy offered to you seem?") and two items measuring affect-focused expectations (e.g., "By the end of the therapy period, how much improvement in your symptoms do you really feel will occur?"). The CEQ applies different rating scales; a 9-point scale ranging from 1 (not at all) to 9 (very much) and a percentage rating scale ranging from 0% (not at all) to 100% (very much) with higher sum scores indicating greater treatment credibility and expectations.

SECONDARY OUTCOMES:
Change from baseline in scores on the Treatment Expectation Questionnaire (TEX-Q) | Baseline; post-Intervention (1 day after baseline, after viewing the intervention videos)
  German version of the Treatment Expectation Questionnaire (TEX-Q), measuring expectations towards psychotherapy in general and towards the process of a psychotherapy (Alberts et al., 2020). Answers are given on a 11-point Likert scale ranging from 0 to 10 (each item has specific anchors with lower anchors always indicating no expected change); The TEX-Q consists of 6 subscales: Treatment benefit (mean item 1,2,3), positive impact (mean item 4,5,6), adverse events (mean item 7,8,9), negative impact (mean item 10,11), process (mean item 12,13), behavioral control (mean item 14,15). TEX-Q overall mean score: mean of all items after inverting items 7-11 with higher scores indicating greater expectations and credibility
Change from baseline in scores on the subscale for treatment expectations of the the generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE) | Baseline; post-Intervention (1 day after baseline, after viewing the intervention videos)
  Prior experiences with psychotherapy and treatment expectations are measured via the generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE), subscale for previous treatment experiences and subscale for treatment expectations (Rief et al., 2021). Answers are provided on a numeric rating scale ranging from 0 to 10 (each item has specific anchors with lower anchors always indicating no expected effects)
Change from baseline in D-Scores on the Single-Category Implicit Associations Test (SC-IAT) | Baseline; post-Intervention (1 day after baseline, after viewing the intervention videos)
  Single-Category Implicit Associations Test (SC-IAT) (Karpinski & Steinman, 2006), measuring implicit associations with psychotherapy. It is a reaction-time task facing the target dimension 'psychotherapy' and the evaluative dimensions 'effective' and 'ineffective'. The strength of the association (D-score) between the target dimension and the evaluative dimension is calculated based on the reaction times. Shorter reaction times indicate a greater associative strength.
Change from baseline in scores on the Credibility and Personal Reaction Scale | Baseline; post-Intervention (1 day after baseline, after viewing the intervention videos)
  Credibility of and personal reactions to psychotherapy are measured via a self-translated German version of the Credibility & Personal Reaction Scales, adapted from Borkovec and Nau (1972) by Addis and Carpenter (1999). This scale also measures intentions to seek therapy.
  Credibility scale: 7 items, answers are provided on a 7-point Likert scale from 1 (not at all) to 7 (extremely).
  Personal Reactions to the Rationales (PRR): 5 items, answers are provided on a 7-point Likert scale from 1 (not at all) to 7 (extremely).
  The total score of the credibility scale ranges from 7 to 49 with higher scores indicating higher credibility ratings, the total PRR score ranges from 5 to 35 with higher scores indicating more positive reactions and higher credibility.
Change from baseline in scores on perceived uncertainty and perceived barriers to psychotherapy | Baseline; post-Intervention (1 day after baseline, after viewing the intervention videos)
  The items used by Kushner and Sher (1989), to assess perceived barriers were translated to German and modified to state "I am uncertain" instead of "I am anxious" (original: Kushner, M. G., & Sher, K. J. (1989). Fear of psychological treatment and its relation to mental health service avoidance. Professional Psychology: Research and Practice, 20(4), 251-257). The scale consists of 3 subscales: therapist responsiveness (5 items), image concerns (4 items), coercion concerns (4 items). Answers are provided on a 5-point scale ranging from 1 (not at all) to 5 (completely) with high scores indicating greater uncertainty. Five items to reflect specific uncertainties (financial concerns, time restrictions, therapist relatability, the therapeutic process, personal ability to complete therapy), that were not covered by the original article, were added. Answers are provided on a 5-point scale ranging from 1 (do not agree) to 5 (agree) with high scores indicating greater uncertainty.
Change from baseline in scores on the Perceived Stigma subscale of the Depression Stigma Scale (DSS) | Baseline; post-Intervention (1 day after baseline, after viewing the intervention videos)
  Public Stigma of depression are measured via the German translation of the Depression Stigma Scale (DSS)(Griffiths et al., 2018), using the Perceived Stigma subscale: 9 items, measuring perceived public stigma of depression. Answers are provided on a 5-point Likert-scale ranging from 0 (completely disagree) to 4 (completely agree); total scores range from 0 to 36 with higher scores indicating greater perceived stigma.
Change from baseline in scores on the Self-Stigma of Depressions Scale (SSDS) | Baseline; post-Intervention (1 day after baseline, after viewing the intervention videos)
  German version of the Self-Stigma of Depressions Scale (SSDS), 16 items measuring anticipated self-stigma for the hypothetical case that one would be suffering from depression (Makowski et al., 2018). The SSDS consists of 3 subscales: self-blame, help-seeking inhibition, social inadequacy Answers on all items are given on a 5-point Likert-scale ranging from 1 (completely disagree) to 5 (completely agree); higher scores indicate higher self-stigma.
Change from baseline in scores on the attitudes towards seeking professional psychological help scale (ATTSPPH-SF) | Baseline; post-Intervention (1 day after baseline, after viewing the intervention videos)
  Attitudes towards seeking professional psychological help (ATTSPPH-SF) - German translation of the short form: 10 items measuring attitudes towards seeking therapy for mental illness (Fischer & Farina, 1995). Answers are given on a 4-point Likert-scale ranging from 0 (disagree) to 3 (agree). The ATTSPPH-SF measures 2 dimensions: openness to seeking professional help for emotional problems (items 1, 3, 5, 6, 7; ) and value and need in seeking professional help (items 2, 4, 8, 9, 10; items inverted: 0 = agree and 3 = disagree). The total score of the scale ranges from 0 to 30 with higher scores indicating a better help-seeking attitude.

OTHER OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Baseline
  Depressive symptoms via the German version of the Patient Health Questionnaire (PHQ-9), 9-item scale (Gräfe et al., 2004). With each item, the PHQ-9 captures one of the nine criteria for major depression posted in the Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) using a 4-point Likert-scale ranging from 0 (not at all) to 3 (almost every day). The total score ranges of 0 to 27, whereby a score of 0 to 4 indicates minimal depressive symptomatology, a score of 5 to 9 mild, a score of 10 to 14 moderate, a score of 15 to 19 moderate to severe, and a total score of 20 to 27 severe depressive symptomatology.
General Self-Efficacy Scale (GSE) | Baseline
  Self-efficacy via the German version of the General Self-Efficacy Scale (GSE), a 10-item scale measuring general self-efficacy (Schwarzer & Jerusalem, 1999). The scale contains 10 items (e.g., "When I am confronted with a problem, I can usually find several solutions"). The answers are presented on a 4-point Likert-scale ranging from 1 (not true at all) to 4 (exactly true) which yields a total score between 10 and 40 with high scores indicating high levels of general self efficacy perceptions.
Empathy on the Interpersonal Reactivity Index (IRI) | Baseline
  Empathy via the German version of the Interpersonal Reactivity Index (IRI), a 16-item scale (Paulus, 2009). Answers are provided on a 5-point rating scale ranging from 1 (never) to 5 (always). Empathy is divided into one cognitive and three emotional components: perspective taking (PT; item 4,10,14,16), fantasy scale (FS; item 2,7,12,15), empathic concern (EC; 1,5,9,11) and personal distress (PD; 3,6,8,13); the general score is determined by the sum value of the individual scales EC, PT and FS (empathy=EC+PT+FS; Paulus, 2012), whereby a higher score indicates higher empathy.
Locus of control perceptions/ "Internale-Externale-Kontrollüberzeugungen-4" (IE-4) | Baseline
  The German 4-item scale IE-4 (Kovaleva et al., 2012) to assess locus of control.
  The IE-4 scale consists of 2 subscales: internal (2 items) and external locus of control (2 items). The 4 items are answered using a 5-point Likert-scale ranging from 1 (strongly disagree) to 5 (strongly agree). The subscale scores are averaged into one score per subscale. The mean subscale values range between 1 and 5 with higher scores indicating higher internal or external locus of control.
Trait uncertainty intolerance/"Unsicherheitsintoleranzfragebogen" (UI-18) | Baseline
  German Uncertainty Intolerance Questionnaire (UI-18), an 18-item scale (Gerlach et al., 2008) to assess trait uncertainty intolerance. The questionnaire assesses three factors ("reduced ability to act due to uncertainty intolerance", "burden due to uncertainty intolerance" and "vigilance due to uncertainty intolerance"). Answers are provided on a 5-point scale ranging from 1 (do not agree) to 5 (agree) with high scores indicating greater uncertainty intolerance.
Cognitive immunization tendencies on the Immunization Scale (IMS) | Baseline
  Cognitive Immunization via the German version of the Immunization Scale (IMS), 31-item scale measuring immunization behavior (Ewen, Rief, & Wilhelm, in progress). The IMS consists of 3 subscales: negative expectations, avoidance, immunization. Answers are provided on a 5-point Likert-scale from 1(do not agree) - 5 (agree) with high scores indicating higher tendencies of negative expectations/avoidance/immunization.
Behavioral proxy variable: Intentions to try a specific technique described in the videos | Post-Intervention (1 day after baseline, after viewing the intervention videos)
  1 item to assess the extent to which participants intend to try a specific technique (emotional writing) presented in each of the videos. Answers are given on a 7-point Likert-scale ranging from 1 (not at all) to 7 (completely).
Warmth and competence ratings of the actors shown in the videos | Post-Intervention (1 day after baseline, directly after viewing the intervention videos)
  Participant perceptions of warmth and competence of actors shown in the videos are measured via the Warmth and Credibility Screener - German translation: 12 items assessing perceived warmth (6 items) and competence (6 items) on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely) with high scores indicating greater ratings of warmth and competence (Seewald & Rief, submitted for publication; English original by Fiske et al., 2002.)
Previous treatment experiences on the subscale for previous treatment experiences of the generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE) | Baseline
  Prior experiences with psychotherapy are measured via the generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE), subscale for previous treatment experiences (Rief et al., 2021). Answers are provided on a numeric rating scale ranging from 0 to 10 (each item has specific anchors with lower anchors always indicating no expected effects)

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Principal Investigator — Department of Clinical Psychology and Psychotherapy, Philipps-University Marburg, Germany, 35032
Locations (1):
- Department of Clinical Psychology and Psychotherapy, Philipps-University Marburg, Marburg, Germany